CLINICAL TRIAL: NCT03647358
Title: Lesion Dosimetry With Iodine-124 in Metastatic Thyroid Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-253
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Carcinoma; Metastatic Thyroid Carcinoma
Keywords: Iodine-124; PET Scan; 18-253
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Positron Emission Tomography Computed Tomography; Iodine-124

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lesion Dosimetry With Iodine-124 (Experimental): Patients will be administered 124I and undergo serial PET imaging consisting of up to 4 individual PET/CT scans. In order to perform a dual exponential fit, 4 scans are needed to obtain the necessary amount of data points required. Lesion dosimetry shall be performed based on the 124I PET scan data through tumor uptake and clearance pharmacokinetics. 10 patients, who sign consent for the sub-study, will be administered an additional tracer diagnostic activity of 124I (4 to 7 mCi). These patients will then undergo additional (up to a maximum of 4) PET scanning during radioiodine therapy at time points matched, if possible, to the days of the pre-therapy 124I dosimetry study.
  Interventions: Device: PET/CT Scan; Drug: Iodine-124

INTERVENTIONS:
Device: PET/CT Scan — Up to four whole-body PET scans (approximately 24, 48, and 120 hours post 124I oral dose) will be performed on one of the GE Discovery 710 or 690 PET scanners.
Drug: Iodine-124 — Patients will receive 0.9 mg injections of rhTSH on two consecutive days. Twenty-four hours after the last injection of rhTSH each patient will receive approximately 5 mCi (range: 4-7 mCi) of 124I orally as a single dose. (If a holiday is present in the work week, 124I can be administered orally on Day 2, if needed).

SUMMARY:
The purpose of this study is to evaluate a new diagnostic imaging test, positron emission tomography (PET), with a different radioactive form of iodine called iodine-124. This form is able to accurately measure the amount of radioactive iodine uptake in the cancer. If the new test determines sufficient radioiodine uptake in the cancer, treatment will continue as usual. However, if the new test shows only low radioiodine uptake, a decision may be made that the benefit from radioiodine therapy is insufficient and that another form of therapy is preferred.

ELIGIBILITY:
Inclusion Criteria:

* Adults with thyroid carcinoma confirmed by pathology.
* Adult thyroid carcinoma patients who have undergone total thyroidectomy
* Adult thyroid carcinoma patients have metastatic disease or suspicion for metastatic disease, or are under a protocol intended to explore re-induction therapy for 131I uptake, and are about to undergo Thyrogen-assisted dosimetry, unless Thyrogen-assisted dosimetry is not required per standard of care.
* The patient and physician are planning to administer 131I for therapy if persistent radioiodine-avid metastases are present.
* All subjects must have measurable disease, documented within the previous six months by ultrasonography (US), MRI, FDG PET/CT, or CT scanning.

Exclusion Criteria:

* Age less than 18 years.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
number of individual lesions response | 1 year
  This will be accomplished using a logistic regression model using lesion as the unit of analysis and adjusting for possible correlation between lesions on the same patient using a random effect at the patient level. by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Grewal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Mauguen A, Grewal RK, Augensen F, Abusamra M, Mahajan S, Jayaprakasam VS, Osborne J, Haque S, Wong BZY, Ghossein RA, Fagin J, Schӧder H, Tuttle RM, Ho A, Humm JL, Larson SM. The use of single-timepoint images to link administered radioiodine activity (MBq) to a prescribed lesion radiation-absorbed dose (cGy): a regression-based prediction interval tool for the management of well-differentiated thyroid cancer patients. Eur J Nucl Med Mol Imaging. 2023 Aug;50(10):2971-2983. doi: 10.1007/s00259-023-06240-1. Epub 2023 May 12. PMID 37171634
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm